CLINICAL TRIAL: NCT03027089
Title: Aspergillus-specific IgG Assays for the Diagnosis of Chronic Pulmonary Aspergillosis (CPA) in Chinese Patients -Multicenter Study
Brief Title: Aspergillus-specific IgG Assays for the Diagnosis of Chronic Pulmonary Aspergillosis (CPA)-Multicenter Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Navy General Hospital, Beijing (Other); Air Force General Hospital of the PLA (Other Government); 307 Hospital of PLA (Other)
Responsible Party: Principal Investigator, Lixin Xie, professor, Chinese PLA General Hospital
Other Study IDs: hr4987
Record Dates: First submitted 2017-01-14; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Pulmonary Aspergillosis
Keywords: Aspergillus-specific IgG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aspergillus-specific IgG assays for the diagnosis of chronic pulmonary aspergillosis (CPA)

DETAILED DESCRIPTION:
chronic pulmonary aspergillosis (CPA) is one of the most refractory pulmonary infectious diseases, and the incidence is increased rapidly in recent years. Serum detection of Aspergillus-specific IgG is considered to be the most reliable method for diagnosing CPA, however, there is no formal report on the appropriate cut-off value for Aspergillus-specific IgG assay in Chinese patients. This study aimed to establish the datum.

Besides aspergillus-specific IgG, there are two other specific antibodies IgM and IgA. IgM is associated with the acute phase of an infection and IgA is associated with mucosal immunity. Their diagnostic values in CPA are still not clear. Meanwhile, whether detection of antibody levels in bronchoalveolar lavage fluid (BALF) could be useful in diagnosis of CPA has not been investigated. In this study, the serum and BALF levels of IgG, IgM and IgA would be detected simultaneously by the commercial available kits.

The investigators will establish the cut-off values of three antibodies by proven CPA patients and negative controls. Then, the cut-off values will be assessed in participants who have a suspected CPA, and the sensitivity, specificity, positive and negative predict value of the antibodies assays will be compared with that of standard diagnostic methods.

After performing the above diagnostic tests, CPA could be diagnosed more accurately and rapidly, so that the antifungal therapy could be evaluated more correctly and timely.

ELIGIBILITY:
Inclusion Criteria:

18 years to 85 years Lesions presented as cavity, nodule，mass or "destroyed lung" caused by fibrosis in CT imaging

Exclusion Criteria:

* seriously immunocompromised patients

  1. Recent history of neutropenia (<0.5 × 109neutrophils/L [<500 neutrophils/mm3] for>10 days) temporally related to the onset of fungal disease
  2. Receipt of an allogeneic stem cell transplant
  3. Prolonged use of corticosteroids (excluding among patients with allergic bronchopulmonary aspergillosis) at a mean minimum dose of 0.3 mg/kg/day of prednisone equivalent for >3 weeks
  4. Treatment with other recognized T cell immunosuppressants, such as cyclosporine, TNF-a blockers, specific monoclonal antibodies (such as alemtuzumab), or nucleoside analogues during the past 90 days
  5. Inherited severe immunodeficiency (such as chronic granulomatous disease or severe combined immunodeficiency)
* antifungal drug use within 3 months of screening
* dropout
* Pregnancy or lactation
* no inform consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects were selected with lesions presented as cavity, nodule，mass or "destroyed lung" caused by fibrosis in CT imaging
Sampling Method: Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The levels of Aspergillus-specific IgG, IgM and IgA in sera and BALF from 560 patients with suspected CPA and 100 healthy blood donors were tested by ELISA assays | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- 301 PLA general hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Denning DW, Cadranel J, Beigelman-Aubry C, Ader F, Chakrabarti A, Blot S, Ullmann AJ, Dimopoulos G, Lange C; European Society for Clinical Microbiology and Infectious Diseases and European Respiratory Society. Chronic pulmonary aspergillosis: rationale and clinical guidelines for diagnosis and management. Eur Respir J. 2016 Jan;47(1):45-68. doi: 10.1183/13993003.00583-2015. PMID 26699723
- [Result] Page ID, Richardson MD, Denning DW. Comparison of six Aspergillus-specific IgG assays for the diagnosis of chronic pulmonary aspergillosis (CPA). J Infect. 2016 Feb;72(2):240-9. doi: 10.1016/j.jinf.2015.11.003. Epub 2015 Dec 8. PMID 26680697
- [Derived] Ma X, Wang K, Zhao X, Liu Y, Li Y, Yu X, Li C, Denning DW, Xie L. Prospective study of the serum Aspergillus-specific IgG, IgA and IgM assays for chronic pulmonary aspergillosis diagnosis. BMC Infect Dis. 2019 Aug 6;19(1):694. doi: 10.1186/s12879-019-4303-x. PMID 31387539